CLINICAL TRIAL: NCT01614028
Title: Total Hip Arthroplasty Using Small Direct Anterior Incision: The Role of Short Femoral Stem
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Other Study IDs: JP2012-01
Record Dates: First submitted 2012-06-04; First posted 2012-06-07 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Total Hip Arthroplasty

ARMS (2):
- Total Hip Arthroplasty using Fitmore femoral stem (Active Comparator)
  Interventions: Procedure: Total Hip Arthoplasty
- Total Hip Arthroplasty using M/L Taper Femoral stem (Active Comparator)
  Interventions: Procedure: Total Hip Arthoplasty

INTERVENTIONS:
Procedure: Total Hip Arthoplasty

SUMMARY:
This study aims to investigate short-term outcomes following the use of two femoral stems used during Total Hip arthoplasty: the Fitmore Femoral stem and the M/L Taper Femoral stem.

ELIGIBILITY:
Inclusion Criteria:

* Patient signed an IRB, study specific informed patient consent.
* Patient is a male or non-pregnant female age 18 years or older at the time of study device implantation.
* Patient has primary diagnosis of non-inflammatory degenerative joint disease.
* Patient is a candidate for primary cementless total hip replacement.
* Patient is willing and able to comply with postoperative scheduled clinical and radiographic evaluations and rehabilitation.

Exclusion Criteria:

* Patient has a Body Mass Index (BMI) > 40 Kg/m2.
* Patient has an active or suspected infection at the time of device implantation.
* Patient is immunologically suppressed.
* Patient requires revision surgery of a previously implanted total hip replacement.
* Patient has a known sensitivity to device materials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Short term hip function | within six weeks post-operative
  Early functional outcome will be measured using the modified Harris Hip score at the first post-operative visit

SECONDARY OUTCOMES:
Short-Term Pain Levels of direct anterior and anterolateral surgical approaches
  Short-term (6 weeks post-op) pain will also be compared between the approach used for the total hip replacement: namely direct anterior and anterolateral using a VAS pain scale

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Rothman Institute at AtlantiCare, Egg Harbor, New Jersey
  - Rothman Institute at Thomas Jefferson University, Philadelphia, Pennsylvania